CLINICAL TRIAL: NCT06346223
Title: Effect of a Single-Session Mindfulness-Based Intervention for Reducing Stress in Family Caregivers of People With Dementia: A Randomized Controlled Trial
Brief Title: Mindfulness-Based Intervention for Family Caregivers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Health and Medical Research Fund (Other Government)
Responsible Party: Principal Investigator, Patrick KOR Pui Kin, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HSEARS20230928006
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Caregiving Stress
Keywords: Family Caregivers; People With Dementia; Mindfulness-Based Intervention
MeSH Terms: conditions — Caregiver Burden | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: A single-blinded, parallel-group, randomized-controlled trial (RCT) design.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness and psychoeducation (Experimental)
  Interventions: Behavioral: Mindfulness and psychoeducation
- Psychoeducation (Active Comparator)
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Mindfulness and psychoeducation — The single-session mindfulness intervention includes a 90-minute group-based session containing different mindfulness practices, psychoeducation and group sharing activities in the single-session mindfulness intervention. A self-practice tool kit will be provided to the participants for home practice 20 minutes daily through an online platform and the participants will be told to develop the practice as a daily habit. All of the teaching contents will be closely related to dementia caregiving and delivered by a mindfulness teacher who has received 40 hours training in dementia caregiving. A weekly mindfulness practice reminder will be sent to the participants through SMS for 8 weeks. The caregivers will also be provided with access to a social media online platform for sharing their practice experience with their classmates online. The interventionist will address their difficulties and challenges via the platform to reinforce skill mastery.
  Arms: Mindfulness and psychoeducation
Behavioral: Psychoeducation — The caregivers in the control group will receive brief education on dementia with the same group size and of the same duration (90-minutes) as the sessions in the intervention arm. The nurse will deliver brief education (15 minutes) on dementia in the session, followed by group sharing and discussion on their daily caregiving experience. The caregivers in the control group will be provided with a toolkit with education materials about the common health problems of older adults and also be given access to a social media platform in which they can communicate and share their caregiving experiences with classmates.
  Arms: Psychoeducation

SUMMARY:
The aim of this study is to investigate the efficiency of a single-session mindfulness-based intervention for reducing stress and promoting psychological health in family caregivers of people with dementia. The single-session mindfulness intervention includes one 90-minute group-based session containing different mindfulness practices, psychoeducation and group sharing activities in the single-session mindfulness intervention. A self-practice tool kit with the teaching materials (e.g., recording of guided mindfulness activities) will be provided to the participants for home practice 20 minutes daily through an online platform and the participants will be told to develop the practice as a daily habit.

Participants will be randomly assigned to receive either the mindfulness intervention combined with psychoeducation or psychoeducation alone. Evaluations will be conducted at baseline (0 weeks), immediately post-intervention (8 weeks), and during a follow-up assessment (6 months). Both groups will complete the same assessments at the same time-points.

DETAILED DESCRIPTION:
The majority of people with dementia receive care from their family members, who assist them with daily activities and managing behavioral problems associated with the illness, such as wandering and agitation. The demanding nature of caregiving tasks, coupled with unpredictable symptoms related to the illness and limited time for other social activities, often leads to high levels of stress among caregivers. By increasing the caregivers' self-awareness in the present moment through the practice of mindfulness, the caregivers tend to step outside their negative experiences and thoughts through a process of decentering, leading to stress reduction. However, considering the growing number of caregivers for people with dementia, there may be insufficient resources to implement intensive mindfulness-based interventions with lengthy durations because most family caregivers are heavily engaged in various caregiving tasks, making a single-session mindfulness-based intervention more suitable for this population compared to a traditional mindfulness program. Although a few pilot studies have demonstrated some preliminary effects of single-session mindfulness-based interventions on promoting mental health, none of these studies focused on family caregivers of individuals with dementia but rather adolescents or adults in general. Further research is necessary to explore the effects of single-session mindfulness-based interventions on reducing stress among family caregivers of individuals with dementia, who experience chronic caregiving stress. Therefore, this study aims to investigate the effectiveness of a single-session mindfulness-based intervention in reducing stress among family caregivers of people with dementia. Additionally, the study will examine other secondary outcomes, such as the impact on the dyadic relationship between caregivers and care-recipients, as well as behavioral and psychological symptoms of dementia.

The target population for this study will be community-dwelling family caregivers of people with dementia. They will be recruited from five elderly centers through the collaboration of two local non-governmental organizations. Interested participants will be assessed for eligibility. After interested and eligible participants provide their consent, they will be randomly assigned to receive either the mindfulness intervention combined with psychoeducation or psychoeducation alone.

The single-session mindfulness intervention includes one 90-minute group-based session containing different mindfulness practices, psychoeducation and group sharing activities in the single-session mindfulness intervention. A self-practice tool kit with the teaching materials (e.g., recording of guided mindfulness activities) will be provided to the participants for home practice 20 minutes daily through an online platform and the participants will be told to develop the practice as a daily habit.

The control group will receive brief education on dementia with the same group size and of the same duration (90-minutes) as the sessions in the intervention arm. The nurse will deliver brief education (15 minutes) on dementia in the session, followed by group sharing and discussion on their daily caregiving experience. The caregivers in the control group will be provided with a toolkit with education materials about the common health problems of older adults and also be given access to a social media platform in which they can communicate and share their caregiving experiences with classmates.

The outcome measures assessed include perceived caregiving stress (primary), depressive symptoms, positive aspect of caregiving, dyadic relationship, trait mindfulness, neuropsychiatric symptoms. Feasibility measures include eligibility and enrollment, attendance rate, adherence to self-practice, and retention rate. Evaluations will be conducted at baseline (0 weeks), immediately post-intervention (8 weeks), and during a follow-up assessment (6 months). Both groups will complete the same assessments at the same time-points.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 or above;
* family caregivers of an individual who has been residing in the community with a confirmed medical diagnosis of any type of dementia (from NGO record or the care-recipients' medical record);
* have been providing care for at least 3 months prior to recruitment with the daily contact of at least 4 hours or more;
* screened positive for caregivers' stress (a summed score of ≥ 25 as measured by the Caregiver Burden Inventory).

Exclusion Criteria:

* have participated in any structured mind-body intervention, or structured psychosocial intervention 6 months prior to recruitment;
* have acute psychiatric condition that are potentially life-threatening or would limit the caregivers' participation in the study (an answer of "yes" to any of the six questions of Columbia Suicide Severity Rating Scale).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Perceived Caregiving Stress in the Family Caregiver | 6 months
  The Perceived Stress Scale (PSS) comprises 10 items rated on a 5-point Likert Scale (0 = never to 4 = very often) to assess perceived stress levels. The total score varies from 0 to 40, with a higher score reflecting more perceived stress. Scores within the ranges of 0-13, 14-26, and 27-40 correspond to low, moderate, and high levels of perceived stress, respectively.

SECONDARY OUTCOMES:
Depressive Symptoms in the Family Caregiver | 6 months
  The Center for Epidemiologic Studies Depression Scale (CESD) comprises 20 items rated on a 4-point Likert scale (0 = rarely or none of the time to 3 = most or almost all the time) to assess the severity of depressive symptoms experienced in the past week. The total score ranges from 0 to 60, with a higher score indicating more severe depressive symptoms. Scores within the ranges of 0-14, 15-21, and 22-60 correspond to low, mild to moderate, and a potential indication of major depression, respectively.
Positive Aspect of Caregiving in the Family Caregiver | 6 months
  The Positive Aspects of Caregiving Scale (PAC) evaluates the perception of positive aspects of caregiving. It consists of 9 items and is rated on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree). A higher score of the PAC suggests a more positive caregiving experience.
Dyadic Relationship Between the Family Caregiver and the Care Recipient | 6 months
  The Dyadic Relationship Scale (DRS) measures the quality of the dyadic relationship between the family caregiver and the care recipient. This scale consists of two versions: the patient version (10 items) and the caregiver version (11 items). Both versions include two subscales: dyadic strain and positive dyadic interaction. They are rated on a 4-point Likert scale (1 = strongly disagree, 4 = strongly agree). Higher scores on each of these scales indicate higher levels of strain and positive interaction, respectively.
Trait Mindfulness in the Family Caregiver | 6 months
  The Five-Facet Mindfulness Questionnaire-Short Form measures trait mindfulness. It consists of 20 items that assess five domains of mindfulness: observing, describing, acting with awareness, nonjudging, and nonreacting. Each domain comprises 4 items and is rated on a 5-point Likert scale (1 = never, 5 = very often). The facet score for each domain is the average of the four items, with higher scores (range = 1-5) indicating higher levels of mindfulness.
Neuropsychiatric Syndromes in the Care Recipient | 6 months
  The Neuropsychiatric Inventory (NPI) measures neuropsychiatric syndromes that occur in Alzheimer's disease and other neurodegenerative disorders. The NPI is administered by the family caregiver and consists of the following domains: Delusions, Hallucinations, Agitation/Aggression, Depression/Dysphoria, Anxiety, Elation/Euphoria, Apathy/Indifference, Disinhibition, Irritability/Lability, and Aberrant Motor Behavior. Each domain is rated based on its frequency (1 = rarely, less than once per week; 4 = very often, once or more per day) and severity (1 = mild, producing little distress in the patient; 3 = severe, very disturbing to the patient and difficult to redirect). A total score can be obtained for each domain by multiplying the frequency and severity ratings. The total score of the NPI is obtained by summing the scores across all domains, with a higher score indicating more severe neuropsychiatric syndromes.
Feasibility of Eligibility and Enrollment | 8 weeks
  Number of eligible participants, and the proportion of those eligible that enrolled will be assessed.
Feasibility of Attendance Rate | 8 weeks
  Number and proportion of attended participants.
Feasibility of Adherence to Self-Practice | 6 months
  The frequency of duration of practicing of mindfulness will be assessed by the number of views and downloads of self-learning materials in an online platform and duration of practice per week in a logbook given to the participants.
Feasibility of Retention Rate | 6 months
  Number and proportion of participants completing all assessments.

REFERENCES:
- [Derived] Kor PPK, Chou KL, Zarit SH, Galante J, Chan WC, Tsang APL, Lai DLL, Cheung DSK, Ho KHM, Liu JYW. Effect of a single-session mindfulness-based intervention for reducing stress in family caregivers of people with dementia: study protocol for a randomized controlled trial. BMC Psychol. 2024 Oct 21;12(1):582. doi: 10.1186/s40359-024-02027-7. PMID 39434193